CLINICAL TRIAL: NCT04288297
Title: Midterm Results After Minimally Invasive Distal Chevron Osteotomy: Comparison of Our Results to the Minimally Invasive Reverdin-Isham Osteotomy From a Systematic Review of the Literature.
Brief Title: Minimally Invasive Distal Chevron in Comparison to the Reverdin-Isham Osteotomy for Hallux Valgus Correction
Status: Completed | Type: Observational
Sponsor: Dr.Gerhard Kaufmann (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor-Investigator, Dr.Gerhard Kaufmann, Dr. Gerhard Kaufmann, Principal investigator and Head of the Orthopaedic and Foot Center Innsbruck, OFZ Innsbruck
Organization: OFZ Innsbruck (Other)
Other Study IDs: 1062/2018
Record Dates: First submitted 2020-02-19; First posted 2020-02-28 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Hallux Valgus and Bunion
MeSH Terms: conditions — Hallux Valgus; Bunion | interventions — austin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- distal minimally invasive distal chevron: The investigators compare the results of a consecutive cohort of patients treated with the above mentioned technique in comparison to the results of patients treated with the minimally invasive Reverdin-Isham technique, presented in literature
  Interventions: Procedure: distal minimally invasive chevron osteotomy

INTERVENTIONS:
Procedure: distal minimally invasive chevron osteotomy — With an electric motor-driven machine the resection of the medial eminence as well as a V-shaped osteotomy was performed in hallux valgus patients. Intraoperative fluoroscopy was used to identify the ideal osteotomy site and to control the Intervention. Fixation of the metatarsal head was achieved with a screw or with a K wire. Residual bone ridges were reamed and bone debris washed out.
  Other Names: austin, v-shaped osteotomy, percutaneous hallux valgus correction

SUMMARY:
This study analyses the Reverdin Isham procedure, which is the most popular minimally invasive surgical hallux valgus correction method and the minimally invasive chevron osteotomy, representing the standard technique of open surgery. It is hypothesized that the two techniques would show significant differences in regard to radiological outcome (Hypothesis 1), clinical outcome (Hypothesis 2) and development of radiological recurrence (Hypothesis 3).

DETAILED DESCRIPTION:
Multiple different surgical techniques have been established for hallux valgus surgery so far, each technique with its unique advantages and limitations. The distal chevron method is widely accepted as a surgical method for correcting mild to moderate hallux valgus deformities. Numerous publications presenting the radiological outcome of this surgical technique and the clinical outcome by means of well established score systems have been published and make this technique, today's benchmark in hallux surgery.

Due to scarring and decreased range of motion of the greater toe joint after open surgery and increasing patients' demands several minimally invasive techniques have been brought to public in the last few years. These techniques claim minor soft tissue damage and reduced surgical time. The efficiency and stability of correction, as well as the clinical outcome of these techniques have been discussed controversially. However, most studies present data from minimally invasive surgery without specific differentiation of the type of surgery and in regard to the clinical and radiological outcome.

Recently a prospective randomized study comparing the open versus the minimally invasive chevron technique has been published presenting data with comparable clinical and radiological outcome.

Given the above-mentioned lack of evidence it was the aim of the study to compare the results of two different minimally invasive techniques. The investigators analyzed the Reverdin Isham procedure, which is known as the technique, that made minimally invasive hallux surgery popular and the minimally invasive chevron osteotomy. It was hypothesized that the two techniques would show significant differences in regard to radiological outcome (Hypothesis 1), clinical outcome (Hypothesis 2) and development of radiological recurrence (Hypothesis 3).

ELIGIBILITY:
Inclusion Criteria:

* patients after minimally invasive distal Chevron osteotomy for hallux valgus deformity with a Minimum follow up of 24 months
* patients with informed written consent for being analyzed
* patients, of whom radiographs are available from preoperative throughout the follow-up time of 24 months

Exclusion Criteria:

* patients under 18 years of age
* pregnant patients, or women below the age of 50 ys, of whom the pregnancy status is not clear
* patients with mental illness or patients, who cannot follow the required postoperative Treatment or controls
* patients, who refuse to participate
* patients, who are assigned to other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A rseries of a cohort of hallux patients treated with the minimally invasive Chevron ostotomy with a Minimum follow-up of 24 months is analyzed retrospectively in regard to the clinical (different clinical scores) and radiological Outcome (radiographic Analysis of defined angles).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
radiological outcome after minimally invasive Chevron osteotomy in comparison to the minimally invasive Reverdin-Isham method presented in literature | change from preoperative to 24 months postoperative (as it is presented in literature)
  radiographic (Hallux valgus angle, Intermetatarsal articular angle and distal metatarsal articular angle measured in grades) with the minimally invasive Chevron osteotomy is evaluated. Data is collected from a consecutive Patient cohort treated at the investigator´s Department. A cohort of more than 50 patients will be assessed.

SECONDARY OUTCOMES:
clinical outcome after minimally invasive Chevron osteotomy in comparison to the minimally invasive Reverdin-Isham method presented in literature | change from preoperative to 24 months postoperative (as it is presented in literature)
  clinical outcome (visual analogue scale- 10 Points maximum, 0 Points Minimum; higher score means worse outcome) with the minimally invasive Chevron osteotomy is evaluated.Data is collected from a consecutive Patient cohort treated at the investigator´s Department. A cohort of more than 50 patients will be assessed.
clinical outcome after minimally invasive Chevron osteotomy in comparison to the minimally invasive Reverdin-Isham method presented in literature | change from preoperative to 24 months postoperative (as it is presented in literature)
  clinical outcome (AOFAS - American Orthopaedic Foot and Ankle Scale- 100 Points maximum, 0 Points Minimum; higher score means better outcome) with the minimally invasive Chevron osteotomy is evaluated.Data is collected from a consecutive Patient cohort treated at the investigator´s Department. A cohort of more than 50 patients will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Gerhard Kaufmann, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vopat BG, Lareau CR, Johnson J, Reinert SE, DiGiovanni CW. Comparative study of scarf and extended chevron osteotomies for correction of hallux valgus. Foot Ankle Spec. 2013 Dec;6(6):409-16. doi: 10.1177/1938640013508431. Epub 2013 Oct 23. PMID 24154993
- [Background] Brogan K, Voller T, Gee C, Borbely T, Palmer S. Third-generation minimally invasive correction of hallux valgus: technique and early outcomes. Int Orthop. 2014 Oct;38(10):2115-21. doi: 10.1007/s00264-014-2500-1. Epub 2014 Aug 17. PMID 25128969
- [Background] Jowett CRJ, Bedi HS. Preliminary Results and Learning Curve of the Minimally Invasive Chevron Akin Operation for Hallux Valgus. J Foot Ankle Surg. 2017 May-Jun;56(3):445-452. doi: 10.1053/j.jfas.2017.01.002. Epub 2017 Feb 22. PMID 28237566
- [Background] Lee M, Walsh J, Smith MM, Ling J, Wines A, Lam P. Hallux Valgus Correction Comparing Percutaneous Chevron/Akin (PECA) and Open Scarf/Akin Osteotomies. Foot Ankle Int. 2017 Aug;38(8):838-846. doi: 10.1177/1071100717704941. Epub 2017 May 5. PMID 28476096
- [Background] Redfern D, Perera AM. Minimally invasive osteotomies. Foot Ankle Clin. 2014 Jun;19(2):181-9. doi: 10.1016/j.fcl.2014.02.002. PMID 24878408
- [Background] Brogan K, Lindisfarne E, Akehurst H, Farook U, Shrier W, Palmer S. Minimally Invasive and Open Distal Chevron Osteotomy for Mild to Moderate Hallux Valgus. Foot Ankle Int. 2016 Nov;37(11):1197-1204. doi: 10.1177/1071100716656440. Epub 2016 Jul 4. PMID 27381179
- [Background] Crespo Romero E, Penuela Candel R, Gomez Gomez S, Arias Arias A, Arcas Ordono A, Galvez Gonzalez J, Crespo Romero R. Percutaneous forefoot surgery for treatment of hallux valgus deformity: an intermediate prospective study. Musculoskelet Surg. 2017 Aug;101(2):167-172. doi: 10.1007/s12306-017-0464-1. Epub 2017 Feb 7. PMID 28168637
- [Background] Maffulli N, Longo UG, Marinozzi A, Denaro V. Hallux valgus: effectiveness and safety of minimally invasive surgery. A systematic review. Br Med Bull. 2011;97:149-67. doi: 10.1093/bmb/ldq027. Epub 2010 Aug 14. PMID 20710024